CLINICAL TRIAL: NCT03412123
Title: Feasibility of the "Lifestyle-integrated Functional Exercise" Concept Delivered in a Group (gLiFE) of Persons Above 70 Years of Age - a Pilot Study
Brief Title: Pilot of a Group-based Program on Lifestyle-integrated Functional Exercise (LiFE) in Older Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); University of Ulm (Other); Universitätsklinikum Hamburg-Eppendorf (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Carl-Philipp Jansen, Post-Doctoral Research Assistant, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01GL1705A
Record Dates: First submitted 2018-01-11; First posted 2018-01-26 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Fall Prevention; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gLiFE pilot group (Experimental)
  Interventions: Behavioral: group lifestyle-integrated functional exercise

INTERVENTIONS:
Behavioral: group lifestyle-integrated functional exercise — Manualized teaching of balance and strength principles and integration of exercises and physical activity into daily routine during 7 sessions in a group of 8 to 10 participants with 2 trainers. The pilot intervention group will undergo the same strength and balance exercises and learn about the same physical activity enhancement strategies as described in the LiFE programme by Clemson et al. (BMJ 2012;345:e4547). However, instead of 7 home visits, gLiFE participants will attend seven group sessions (1 session/week). In these, LiFE contents are adapted to the group setting and enhanced by health psychological and behaviour change strategies fitting to the social structure and modalities of a group.

SUMMARY:
This feasibility pilot is part of the project "LiFE-is-LiFE" (2017-2020). It is based on the Lifestyle-Integrated Functional Exercise (LiFE) program by Clemson et al., which has proven effective in improving strength, balance, and physical activity while simultaneously reducing falls in older people via incorporating exercises in recurring daily tasks. However, implementing the original LiFE program includes high financial requirements and human resources. Therefore, LiFE-is-LiFE investigates whether implementing LiFE in groups (gLiFE) is not inferior to the original, individually delivered LiFE in terms of reducing falls per physical activity. In this pilot study, we evaluate our conception of gLiFE for large-scale use in the subsequent, larger LiFE-is-LiFE trial.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling
* Aged 70+

Exclusion Criteria:

* Cognitive impairment
* Neurological condition which severely influences gait and mobility
* Severe visual impairment
* Inability to ambulate independently
* Significant lung disease or chronic heart failure or any other unstable or terminal illness that would preclude the planned exercises

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Adherence of the participants to LiFE activities | Change from the first of 7 intervention sessions (i.e., at week 1) at the end of the intervention period (i.e., week 7)
  Measured using the Exercise Adherence Rating Scale (EARS)
Evaluation of the intervention and its components | at the end of the intervention period (i.e., week 7)
  Rating of helpfulness (5-point Likert scale), safety (5-point Likert scale), level of difficulty (5-point Likert scale), and adaptability (5-point Likert scale)
Participants' views on the gLiFE program | at the end of the intervention period (i.e., week 7)
  Participants' views on:
  1. planning and engaging in gLiFE activities
  2. the gLiFE manual
  3. support from the trainers
  4. their ideas for improving the program
  5. the group format

SECONDARY OUTCOMES:
Functional performance | Change from baseline (i.e., before the first session) at the end of the intervention period (i.e., week 7)
  Timed up-and-go test (measured in seconds; shorter time represents better performance)
Motor performance (balance) | Change from baseline (i.e., before the first session) at the end of the intervention period (i.e., week 7)
  8 Level balance scale (measured in accomplished levels; higher level represents better performance)
Motor performance (strength) | Change from baseline (i.e., before the first session) at the end of the intervention period (i.e., week 7)
  5-chair rise (measured in seconds; shorter time represents better performance)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schwenk, PhD, Principal Investigator — Heidelberg University; Clemens Becker, MD, Study Chair — Robert Bosch Medizinische Gesellschaft mbH
Locations (1):
- Heidelberg University, Network Aging Research, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kramer F, Labudek S, Jansen CP, Nerz C, Fleig L, Clemson L, Becker C, Schwenk M. Development of a conceptual framework for a group-based format of the Lifestyle-integrated Functional Exercise (gLiFE) programme and its initial feasibility testing. Pilot Feasibility Stud. 2020 Jan 22;6:6. doi: 10.1186/s40814-019-0539-x. eCollection 2020. PMID 31993213
- See also: Website of the overall LiFE-is-LiFE trial — http://www.life-alltagsuebungen.de
- See also: Project website as part of the overall working group's website — http://www.nar.uni-heidelberg.de/juniorforscher/ng_schwenk/lifeislife.html